CLINICAL TRIAL: NCT05761990
Title: Effects Of A Novel Stretching Versus Post Isometric Relaxation Techniques On Shoulder Pain, Range Of Motion And Disability In Overhead Athletes With Glenohumeral Internal Rotation Deficits
Brief Title: Novel Stretching Versus Post Isometric Relaxation Techniques On Shoulder Disability In Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0412
Record Dates: First submitted 2022-11-24; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Glenohumeral Internal Rotation Deficit
Keywords: range of motion,pain,shoulder,stretching

STUDY DESIGN:
Intervention Model Description: POSTERIOR ISOMETRIC TECHNIQUES
  * For 5 to 10 seconds, a submaximal (10-20%) hypertonic muscle contraction is carried out away from the barrier while resistance is supplied in the other side.
  * The individual is told to relax while breathing after the isometric contraction. After then, until the next barrier is reached, a gentle stretch is employed to pick up the slack.
  NOVEL STRETCHING TECHNIQUE The NS will be performed in a supine posture for Group B participants. Participants will be instructed to open their knees while wearing a resistance band around their knees. Participant will be instructed to bridge as high as he can while keeping his shoulders 90 ° abducted and his elbows 90 ° flexed. By lifting the body weight upward, the bridging motion pins the scapula's medial border against the thorax without immediately squeezing or constricting the posterior shoulder bones.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POST ISOMTERIC RELAXATION TECHNIQUES (Experimental): Participants in Group A will instruct to perform the PIR techniques
  These steps are taken when using the PIR approach:
  * Stretching the hypertonic muscle to the point when movement resistance is initially felt or just past the point of discomfort.
  * For 5 to 10 seconds, a submaximal (10-20%) hypertonic muscle contraction is carried out away from the barrier while resistance is supplied in the other side. To help with this, the individual should breathe in.
  * The individual is told to relax while breathing after the isometric contraction. After then, until the next barrier is reached, a gentle stretch is employed to pick up the slack.
  * Starting with this new barrier, the procedure is carried out two or three more times.
  Interventions: Other: POST ISOMTERIC RELAXATION TECHNIQUE
- NOVEL STRETCHING (Experimental): The NS will be performed in a supine posture for Group B participants. Participants will be instructed to open their knees while wearing a resistance band around their knees. Participant will be instructed to bridge as high as he can while keeping his shoulders 90 ° abducted and his elbows 90 ° flexed. By lifting the body weight upward, the bridging motion pins the scapula's medial border against the thorax without immediately squeezing or constricting the posterior shoulder bones. This position is thought to provide more flexibility of mobility while causing less discomfort. The subjects were instructed to hold this position while tightening or "squeezing" their gluteal muscles. They were also instructed to stretch by jerkily turning their shoulders inward as far as possible. Using the second hand, the stretch was pushed forward to the point of mild discomfort while contraction was maintained.
  Interventions: Other: NOVEL STRETCHING

INTERVENTIONS:
Other: POST ISOMTERIC RELAXATION TECHNIQUE — POST ISOMETRIC RELAXATION TECHNIQUES
  * Stretching the hypertonic muscle to the point when movement resistance is initially felt or just past the point of discomfort.
  * For 5 to 10 seconds, a submaximal (10-20%) hypertonic muscle contraction is carried out away from the barrier while resistance is supplied in the other side. To help with this, the individual should breathe in.
  * The individual is told to relax while breathing after the isometric contraction. After then, until the next barrier is reached, a gentle stretch is employed to pick up the slack.
  * Starting with this new barrier, the procedure is carried out two or three more times.
  Arms: POST ISOMTERIC RELAXATION TECHNIQUES
Other: NOVEL STRETCHING — NOVEL STRETCHING The NS will be performed in a supine posture for Group B participants. Participants will be instructed to open their knees while wearing a resistance band around their knees. Participant will be instructed to bridge as high as he can while keeping his shoulders 90 ° abducted and his elbows 90 ° flexed. By lifting the body weight upward, the bridging motion pins the scapula's medial border against the thorax without immediately squeezing or constricting the posterior shoulder bones. This position is thought to provide more flexibility of mobility while causing less discomfort. The subjects were instructed to hold this position while tightening or "squeezing" their gluteal muscles. They were also instructed to stretch by jerkily turning their shoulders inward as far as possible. Using the second hand, the stretch was pushed forward to the point of mild discomfort while contraction was maintained.
  Arms: NOVEL STRETCHING

SUMMARY:
It was a randomized control trial in which thirty (30) participants having GRID, age between 20-40 years were randomly allocated into two groups i-e NS (Novel stretching) Group (30) and PIR (posterior isometric relaxation techniques) Group (30), February 2022 to March 2022.PIR group received the posterior isometric relaxation techniques (three times a week for one month) and NS group received the Novel stretching (three times a week for one month). IR ROM was measured with a goniometer while pain was measured with Numeric Pain Rating Scale intervention and disability of arm, shoulder and hand was measured with DASH score before, immediately, and at week 4 post intervention.

ELIGIBILITY:
Inclusion Criteria:

* Male and female
* Between the ages of 18 and 40
* Athletes with glenohumeral internal deficit
* Basketball, tennis, javelin, squash, swimmers, volleyball, and weightlifter
* participated in local and regional sporting events
* showed a 10° or higher variation in Internal rotation range of motion between shoulders (dominant versus non-dominant)

Exclusion Criteria:

* Footballer, cricketer, and hockey player
* Recovering from extensive shoulder and elbow surgery that was performed three months ago.
* presently undergoing medical intervention for the shoulder
* Suffer from a life-threatening illness

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-07-17 (Actual); Primary Completion 2022-09-17 (Actual); Study Completion 2022-09-17 (Actual)

PRIMARY OUTCOMES:
numeric pain rating scale | 4weeks
  A respondent uses the Numeric pain rating scale, a numerical variant of the visual analogue scale (VAS), to select a whole number (0-10 integers) that best captures the severity of their pain.
RANGE OF MOTION | 4 weeks
  The ROM is measured by GONIOMETER
Disability of arm,shoulder and hand score | 4 weeks
  The DASH is a 30-item questionnaire that offers response options using 5-point Likert scales. Scores vary from 0 (no disability) to 100 (complete disability) (most severe disability). This score was created to help patients with any upper-limb musculoskeletal problem

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Sanaullah, MS, Principal Investigator — Riphah International University
Locations (1):
- Muhammad Sulaman, Multan Khurd, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lacheta L, Horan MP, Nolte PC, Goldenberg BT, Dekker TJ, Millett PJ. SLAP Repair Versus Subpectoral Biceps Tenodesis for Isolated SLAP Type 2 Lesions in Overhead Athletes Younger Than 35 Years: Comparison of Minimum 2-Year Outcomes. Orthop J Sports Med. 2022 Jun 21;10(6):23259671221105239. doi: 10.1177/23259671221105239. eCollection 2022 Jun. PMID 35757237
- [Background] Jung JW, Kim YK. Scapular Dyskinesis in Elite Boxers with Neck Disability and Shoulder Malfunction. Medicina (Kaunas). 2021 Dec 9;57(12):1347. doi: 10.3390/medicina57121347. PMID 34946291